CLINICAL TRIAL: NCT06894511
Title: A Phase II, Open-label, Multi-Center, Randomized Study Comparing the Combination of Lutetium (177Lu) Vipivotide Tetraxetan (AAA617) and Androgen Receptor Pathway Inhibitor (ARPI) vs. Lutetium (177Lu) Vipivotide Tetraxetan (AAA617) in First-line Treatment of Patients With Prostate-Specific Membrane Antigen (PSMA)-Positive Progressive Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: An Open-label Study Comparing Lutetium (177Lu) Vipivotide Tetraxetan (AAA617) in Combination With ARPI Versus AAA617 in PSMA Positive First-line mCRPC
Acronym: PSMAndARPI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAA617B1US01
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration Resistant Prostate Cancer (mCRPC)
Keywords: Prostate-specific membrane antigen (PSMA); lutetium (177Lu) vipivotide tetraxetan (AAA617); Androgen Receptor Pathway Inhibitors (ARPI); Enzalutamide; Abiraterone; Apalutamide; Darolutamide; metastatic Castration Resistant Prostate Cancer (mCRPC)
MeSH Terms: interventions — Lutetium; Lutetium-177; Pluvicto

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: AAA617 and ARPI (Experimental): AAA617 and ARPI (Enzalutamide, Abiraterone):
  * AAA617 will be administered once every 6 weeks (1 cycle) for a planned 6 cycles.
  * ARPI will be administered from 14 days (+ 7 days) before first dose of AAA617 until participant is no longer clinically benefiting, or experiences unacceptable toxicity or if investigator determines that the patient should discontinue ARPI.
  Interventions: Drug: AAA617; Drug: ARPI: Abiraterone; Drug: ARPI: Enzalutamide
- Arm B: AAA617 alone (Active Comparator): AAA617 alone: Control Arm B participants will receive a dose of AAA617 which will be administered once every 6 weeks (1 cycle) for a planned 6 cycles.
  Interventions: Drug: AAA617

INTERVENTIONS:
Drug: AAA617 — Dose formulation: open-label vial
  Dose level: 7.4 GBq (200 mCi) ± 10% Once, every 6 weeks for 6 cycles, intravenous administration
  Other Names: lutetium (177Lu) vipivotide tetraxetan; [177Lu]Lu-PSMA-617; 177Lu-PSMA-617
Drug: ARPI: Abiraterone — Dose formulation: tablet/capsule
  Dose level: 160 mg (four 40 mg or two 80 mg soft capsules) as a single daily dose, oral administration
  Arms: Arm A: AAA617 and ARPI
Drug: ARPI: Enzalutamide — Dose formulation: tablet
  Dose level: 1000 mg daily (two 500 mg tablets or four 250 mg tablets as a single daily dose together with 5 mg oral prednisone 2 times a day, oral administration
  Arms: Arm A: AAA617 and ARPI

SUMMARY:
The purpose of this study is to assess whether the combination of AAA617 (administered for 6 cycles at a dose of 7.4 GBq (200 mCi) +/- 10%) and ARPI improves radiographic progression-free survival (rPFS) or time to death compared to AAA617 alone in PSMA-positive mCRPC patients who were previously treated and progressed on ARPI in the biochemical recurrence (BCR)-non metastatic hormone sensitive prostate cancer (mHSPC), mHSPC, or non-metastatic Castration Resistant Prostate Cancer (nmCRPC) setting and have not previously received a taxane-containing regimen in the castrate resistant prostate cancer (CRPC) setting.

DETAILED DESCRIPTION:
This prospective, open-label, multi-center, randomized phase II study will enroll adult participants with PSMA PET positive mCRPC who were previously treated and progressed on ARPI in the BCR-non mHSPC, mHSPC, or nmCRPC setting and have not previously received a taxane-containing regimen in the CRPC setting. A PSMA PET/ computed tomography (CT) scan will be done at Screening to confirm PSMA positive disease. This is a United States-based study.

Approximately 420 eligible participants will be randomized in a 1:1 ratio to one of the two treatment arms (Arm A: AAA617+ARPI vs Arm B: AAA617). The primary objective of the study is to evaluate the rPFS response in participants with metastatic CRPC, assessed by conventional imaging, treated with AAA617 in combination with ARPI and AAA617 alone. Best Supportive Care (BSC) will be allowed in both arms at the discretion of the investigator and includes available care for the eligible participants according to best institutional practice for mCRPC. Androgen deprivation therapy (ADT) is required in both arms.

A total of approximately 420 eligible participants will be randomized in a 1:1 ratio into one of two treatment arms. Participants in Arm A will receive AAA617 in combination with ARPI, while those in Arm B will receive AAA617 alone. Randomization will be stratified by type of prior ARPI (abiraterone vs other [enzalutamide, apalutamide, or darolutamide]) and by setting of prior ARPI (mHSPC without docetaxel vs mHSPC with docetaxel vs others [BCR-non mHSPC or nmCRPC setting]).

The study duration is approximately 3.5 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have an ECOG performance status of 0 to 2.
* Participants must have histopathological, and/or cytological confirmation of adenocarcinoma of the prostate.
* Participants must have PSMA PET positive disease using FDA approved PSMA-imaging approved agents, and eligible as determined by the sponsor's central reading rules.
* Participants must have a castrate level of serum/plasma testosterone (< 50 ng/dL or < 1.7 nmol/L).
* Newly diagnosed mCRPC participants who must have progression on prior ARPI in the BCR-non mHSPC, mHSPC, or nmCRPC setting.
* Participants must have progressed only once on prior second-generation ARPI (abiraterone, enzalutamide, darolutamide, or apalutamide). First generation androgen receptor inhibitor therapy (e.g. bicalutamide) is allowed but not considered as prior ARPI therapy (second generation ARPI must be the most recent therapy received).
* Participant must have been diagnosed with mCRPC with documented progressive disease after having been previously treated with ARPI in the BCR-non mHSPC, mHSPC, or nmCRPC setting as their last treatment (and did not progress on more than one ARPI), based on at least 1 of the following criteria:

  * Serum/plasma PSA progression is defined as 2 increases in PSA measured at least 1 week apart. The minimal start value is 2.0 ng/mL; 1.0 ng/mL is the minimal starting value if confirmed rise in PSA is the only indication of progression as per PCWG3 guidelines.
  * Soft-tissue progression defined [PCWG3-modified RECIST v1.1 (Eisenhauer et al 2009, Scher et al 2016)].
  * Progression of bone disease: 2 new lesions; only positivity on the bone scan defines metastatic disease to bone (PCWG3 criteria [Scher et al 2016]).
* Participants must have ≥ 1 metastatic lesion by conventional imaging that is present at Screening/Baseline CT, MRI, or bone scan imaging obtained ≤ 28 days (about 4 weeks) prior to randomization.
* Participants must have adequate organ function:

Bone marrow reserve

* Absolute Neutrophil Count (ANC) ≥ 1.5 × 109/L
* Platelets ≥ 100 × 109/L
* Hemoglobin ≥ 9 g/dL Hepatic
* Total bilirubin < 2 × the institutional upper limit of normal (ULN). For participants with known Gilbert's Syndrome ≤ 3 × ULN is permitted.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 3.0 × ULN OR ≤ 5.0 × ULN for participants with liver metastases
* Albumin ≥ 2.5 g/dL Renal
* eGFR ≥ 50 mL/min/1.73m2 using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.

Exclusion Criteria:

* Previous treatment with any of the following within 6 weeks of randomization: Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-body irradiation, and Lu-DOTA radioligand therapy.
* Previous PSMA-imaging RLT
* Previous treatment with taxane-based chemotherapy at mCRPC settings. Taxane exposure is allowed in the mHSPC setting if more than 12 months have elapsed since the completion of this therapy.
* Participants with a history of CNS metastases who are neurologically unstable, symptomatic, or receiving corticosteroids for the purpose of maintaining neurologic integrity.
* Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression.
* Participant with known or suspected deleterious germline or somatic homologous recombination repair gene-mutated mCRPC, who is considered appropriate for treatment with PARP inhibitor according to the judgment of the investigator.
* History of myocardial infarction, angina pectoris, or coronary artery bypass graft (CABG) within 6 months prior to ICF signature and/or clinically active significant cardiac disease
* Concurrent serious acute or chronic nephropathy as determined by the principal investigator.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2025-09-11 (Actual); Primary Completion 2029-04-09 (Estimated); Study Completion 2029-04-09 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression Free Survival (rPFS) | From date of randomization to date of first documented radiographic disease progression or death due to any cause, whichever occurs first, up to approximately 24 months
  Time to radiographic disease progression or death due to any cause as assessed by Blinded Independent Central review (BICR) using conventional imaging and PCWG3-modified RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization to date of death due to any cause, up to approximately 24 months
  Time to death due to any cause
Progression-free survival (PFS) | From date of randomization to date of first documented progression or death from any cause, whichever occurs first, up to approximately 24 months
  Time to first documented progression or death from any cause per investigator's assessment (radiographic, clinical, or Prostate Specific Antigen (PSA) progression).
Secondary PFS2 | From date of randomization to first documented progression or death from any cause, whichever occurs first, for up to approximately 24 months
  Time to first documented progression or death from any cause by investigator's assessment (radiographic progression, clinical progression, PSA progression) on next line of therapy
Overall response rate (ORR) | From date of randomization to date of first documented progression or death due to any cause, whichever occurs first, up to approximately 24 months
  The proportion of participants with best overall response (BOR) of confirmed complete response (CR) or partial response (PR) in soft tissue based on tumor response data per BICR assessment and according to PCWG3-modified RECIST v1.1, in the absence of bone progression as per PCWG3-modified RECIST v1.1. Additionally, ORR in soft tissue only according to PCWG3-modified RECIST v1.1 will be analyzed.
Disease control rate (DCR) | From date of randomization to date of first documented progression or death due to any cause, whichever occurs first, up to approximately 24 months
  The percentage of participants with best overall response (BOR) of confirmed complete response (CR), partial response (PR), stable disease (SD) or Non-CR/Non-progressive disease (PD) in soft tissue based on tumor response data per BICR assessment and according to PCWG3-modified RECIST v1.1, in the absence of bone progression as per PCWG3-modified RECIST v1.1
Duration of response (DoR) | From date of first documented response (CR or PR) and date of first documented radiographic progression in soft tissue or death due to any cause, whichever occurs first, up to approximately 24 months
  Time between the date of first documented response and the date of first documented radiographic progression or death due to any cause, according to PCWG3-modified RECIST v1.1, in the absence of bone progression as per PCWG3-modified, based on tumor response data per BICR.
Biochemical response by prostate specific antigen (PSA50 and PSA90) response rate | From baseline to date of first documented progression or death due to any cause, whichever occurs first, up to approximately 24 months
  The percentage of participants who achieved ≥ 50% and ≥ 90% decrease in PSA from baseline, respectively, that is confirmed by a second PSA measurement ≥4 weeks
Time of first symptomatic skeletal event (TTSSE) | From date of randomization to date of first symptomatic skeletal event or death due to any cause, whichever occurs first, up to approximately 24 months
  Time to first new symptomatic skeletal event (symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, or requirement for radiation therapy to relieve bone pain) or death due to any cause, whichever occurs first, up to approximately 24 months.
Time of first radiographic soft tissue progression (TTSTP) | From date of randomization to date of radiographic soft tissue progression or death due to any cause, whichever occurs first, up to approximately 24 months
  Time to radiographic soft tissue progression per soft tissue rules of PCWG3-modified RECIST v1.1 as assessed by BICR.
Time to initiation of cytotoxic chemotherapy | From date of randomization to date of first documented dose of new cytotoxic chemotherapy or death due to any cause, whichever occurs first, up to approximately 24 months
  Time to first documented dose of new cytotoxic chemotherapy being administered to the participant.
Brief Pain Inventory-Short Form (BPI-SF) | From date of randomization to date of worsening of worst pain intensity, up to approximately 24 months
  Time to worsening of worst pain intensity or death due to any cause. Worsening of worst pain intensity is defined as first occurring 1) an increase of worsening threshold compared to baseline, 2) clinical disease progression or 3) death.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United States (14):
  - Cancer And Blood Spclsts of AZ, Casa Grande, Arizona
  - Arizona Center for Cancer Care, Gilbert, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Univ Of Color Anschutz Med Center, Aurora, Colorado
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - East Jefferson Hospital, Metairie, Louisiana
  - Urology Cancer Center PC, Omaha, Nebraska
  - Northwest Cancer Specialists, Portland, Oregon
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology P A, Bedford, Texas
  - Urology Austin, Lakeway, Texas
  - Urology San Antonio, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com